CLINICAL TRIAL: NCT00492102
Title: Pharmacokinetics of Montelukast in Very Low Birthweight (VLBW) Preterm Infants
Brief Title: Montelukast in Very Low Birthweight Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCHMC IRB# 05-05-22; TriHealth IRB# 05037-0505 (Other: TriHealth IRB)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: pharmacokinetics; Montelukast; bronchopulmonary dysplasia; Pharmacokinetics of Montelukast
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Nine VLBW pre-term infants older than 7 days will be enrolled in the study and receive one oral dose of Montelukast based on weight. Two blood samples will be obtained from each infant within 24 hours of the drug administration and plasma Montelukast levels will be determined.
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — One oral dose of Montelukast 0.15mg (infants weighing 500-1000gm) or 0.2mg (infants weighing >1000gm). Two blood samples will be obtained from each infant within 24 hours of the drug administration and plasma Montelukast levels will be determined.
  Other Names: Singulair

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (PK) of montelukast (Singulair) in very low birth weight (VLBW) infants at risk for developing bronchopulmonary dysplasia (the need for supplemental oxygen). The investigators' long-term hypothesis is that inhibition of leukotriene signaling in the VLBW preterm lung will decrease inflammation, remodeling and the incidence of bronchopulmonary dysplasia (BPD).

DETAILED DESCRIPTION:
This study proposal will determine the pharmacokinetics (PK) of montelukast (cysteinyl leukotriene receptor-1 or CysLT1 inhibitor) in very low birth weight (VLBW) infants between 500 - 1500g birth weight at risk for developing bronchopulmonary dysplasia (BPD). Montelukast (Singulair) is a FDA approved specific CysLT1 antagonist widely used clinically in the prophylaxis of asthma in children older than 12 months of age and blocks leukotriene signaling in the lung. BPD shares some pathogenic mechanisms with asthma, however Cysteinyl LT receptor blockade has not been studied in preterm infants. Montelukast is metabolized by the cytochrome P450 system which is immature in the preterm infant and hence the need for this study. The investigators' long-term hypothesis is that inhibition of leukotriene signaling in the VLBW preterm lung will decrease inflammation, remodeling and the incidence of BPD. The data will be used to design future efficacy trials of Montelukast in the prevention of bronchopulmonary dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* VLBW infants between 500 - 1500 gm birth-weight born at Good Samaritan Hospital, Cincinnati, tolerating oral feeds equal to or more than 75 ml/kg/day and older than 7 days

Exclusion Criteria:

* Infants diagnosed with congenital malformations.
* Infants with an acute life threatening illness.
* Grade III or IV intra-ventricular hemorrhage.
* Patent ductus arteriosus being treated with indomethacin.
* Oral feedings are contra-indicated.
* Parents refuse consent.
* Attending physician does not wish the infant to be enrolled in the study.
* Infants with known hepatitis or HIV.
* Infants enrolled in any study using an investigational drug.

Min Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determine the pharmacokinetics of Montelukast in very low birth weight infants between 500 - 1500 g birth weight at risk for developing bronchopulmonary dysplasia | 72 hours
Evaluate the preliminary safety of montelukast in pre-term neonates (single dose). | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Suhas Kallapur, MD, Principal Investigator — CCHMC/Good Samaritan
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States